CLINICAL TRIAL: NCT06614634
Title: Comparison of Center-Based and Tele Cardiac Rehabilitation on Functional Capacity, Quality of Life, and Fear of Activity in Coronary Artery Disease: A Patient-Preferred, Controlled, Prospective Study
Brief Title: Comparison of Conventional and Tele-cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Levent Karataş, M.D., Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Cardiac telerehab
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease; Cardiac Rehabilitation; Telecardiac Rehabilitation; Aerobic Exercise
Keywords: Cardiac rehabilitation; Telerehabilitation; Coronary artery disease; Tele-cardiac rehabilitation; Fear of activity
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients with coronary artery disease who met the inclusion criteria were allocated into hospital-based and tele-cardiac rehabilitation groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-cardiac rehabilitation group (Experimental): Patients in the tele-cardiac rehabilitation group initially underwent a similar trial exercise session as those in the hospital-based rehabilitation group. During this session, patients were informed about exercise duration and intensity, using the heart rate monitor (Polar H9) and elastic bands, and transferring data to the web application (Polar Flow web). Subsequently, patients were instructed to perform aerobic and strengthening exercises at home/outdoors at least 3 days a week for four weeks. During the program, the researcher called them once a week for reinforcement. Phone calls included symptom inquiry and encouraging feedback regarding exercise parameters recorded on the Polar H9 website in the previous week. In the second week, patients underwent an interim exercise session under supervision in our CPR unit and a similar face-to-face interview was conducted. The program was concluded at the end of four weeks.
  Interventions: Other: Remotely supervised exercise at home or outdoors; Behavioral: Cardiovascular risk modification; Other: Phone calls with reinforcement feedback
- Hospital-based rehabilitation group (Active Comparator): Participants in the hospital-based rehabilitation group performed aerobic and strengthening exercises under the supervision of a physiotherapist/nurse/research doctor three days a week for four weeks in the cardiopulmonary rehabilitation unit. Aerobic exercise included 30-minute treadmill walking at 60-80% of the peak VO2 value obtained in the cardiopulmonary exercise test. After the end of the aerobic exercise, upper and lower extremity muscle strengthening exercises were performed with warm-up and cool-down periods using medium-tension elastic bands under the supervision of a physiotherapist. At the end of four weeks, the program was terminated and a follow-up evaluation was conducted.
  Interventions: Other: Hospital-based exercise program; Behavioral: Cardiovascular risk modification

INTERVENTIONS:
Other: Remotely supervised exercise at home or outdoors — Aerobic and strengthening exercise program at home/outdoors at least three days a week for four weeks using a Polar H9 heart rate monitor and elastic band.
  Arms: Tele-cardiac rehabilitation group
Other: Hospital-based exercise program — The aerobic and strengthening exercise program three days a week for four weeks under supervision in our cardiopulmonary rehabilitation unit.
  Arms: Hospital-based rehabilitation group
Behavioral: Cardiovascular risk modification — Psychosocial support for physical activity counselling, heart-healthy diet, referral for smoking cessation and stress management.
Other: Phone calls with reinforcement feedback — Calls once a week that include symptom inquiries and encouraging feedback on exercise logs.
  Arms: Tele-cardiac rehabilitation group

SUMMARY:
This study aimed to compare the effects of tele-cardiac rehabilitation (TCR) and hospital-based cardiac rehabilitation (HBCR) on functional capacity (maximum oxygen consumption), fear of activity and quality of life in patients with coronary artery disease. CAD). The rehabilitation program included patient-specific aerobic and peripheral muscle strengthening exercises for four weeks and 3 sessions per week. While the HBCR group performed the exercise program under supervision in the cardiac rehabilitation (CR) unit, the TCR group performed the exercise program at home/outdoors using a Polar H9 heart rate monitor and elastic band.

DETAILED DESCRIPTION:
This prospective, patient-preference, controlled study aimed to investigate the comparative effects of tele-cardiac rehabilitation (TCR) and hospital-based cardiac rehabilitation (HBCR) on functional capacity, fear of activity, and quality of life in patients with coronary artery disease (CAD). The study was conducted between February 2022 and May 2024 at the university's Physical Medicine and Rehabilitation Department. Patients were enrolled based on specific inclusion and exclusion criteria, including stable CAD and adequate technological access for TCR participation. The study design allowed participants to choose between TCR and HBCR after receiving information about both programs, reflecting real-life clinical decision-making scenarios.

Both rehabilitation programs lasted for four weeks, with three exercise sessions per week. In the HBCR group, patients underwent supervised exercise sessions in the cardiac rehabilitation (CR) unit, including individualized aerobic and resistance training. Aerobic exercises were based on the patient's peak VO2 from a baseline cardiopulmonary exercise test (CPET), aiming to achieve 60-80% of the maximum heart rate. Resistance training involved the use of elastic bands targeting major muscle groups, with a progressive increase in repetitions based on patient tolerance.

The TCR group received a home-based exercise program that included aerobic and resistance training. Aerobic exercises, such as walking, were performed for 30 minutes, three times a week, monitored via a Polar H9 heart rate device. Patients were instructed to maintain heart rates within the same range as the HBCR group. Resistance exercises were similar to those in the HBCR group, using elastic bands provided at the beginning of the study. Weekly remote follow-ups were conducted via phone calls to assess adherence, review heart rate data, and provide encouragement.

Initial and final evaluations included the CPET, the Coronary Artery Disease-Specific Activity Fear Scale (AKKOR-KAH), and the WHOQOL-BREF Quality of Life Questionnaire. Outcome measures assessed changes in peak oxygen consumption (VO2 max), exercise capacity, quality of life, and fear of activity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of clinically stable coronary artery disease (CAD), defined as stable angina pectoris, a history of myocardial infarction, history of percutaneous coronary intervention, or coronary artery bypass graft surgery.
* Classified as having a low to moderate risk of experiencing a new cardiac event, according to established risk stratification guidelines.
* Possession of a smartphone and reliable internet access at home to facilitate participation in telehealth interventions.

Exclusion Criteria:

* Presence of severe ventricular arrhythmias during low to moderate exercise intensity or a documented history of myocardial ischemia, unstable angina, or abnormal exercise test results during initial evaluation.
* Presence of a pacemaker or implantable cardioverter-defibrillator that may interfere with study protocols.
* Hospitalization for any cardiac condition within the last 6 weeks prior to enrollment.
* Evidence of residual coronary artery stenosis necessitating revascularization procedures.
* Classification of heart failure as New York Heart Association (NYHA) Class IV, indicating severe functional limitations.
* Diagnosis of untreated malignancy that could affect participation and outcomes.
* Presence of orthopedic, neurological, or psychiatric disorders that may hinder assessment or engagement in prescribed exercise regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
World Health Organization Quality of Life Scale-BREF score | From enrollment day to the end of the rehabilitation program at 4 weeks
  This scale is used for a brief assessment of the quality of life in routine clinical practice, large-scale epidemiological studies, or clinical trials. It comprises 27 questions that evaluate general health status, physical health, psychological status, social relations and environmental issues sub-titles. Each question receives an answer corresponding to 1-5 points. The percentages of the scores obtained from each sub-title allow us to make a quantitative interpretation of domains of the quality of life. Increased scores represent higher life quality.
Maximum oxygen consumption (VO₂ max) | From enrollment day to the end of the rehabilitation program at 4 weeks
  It is the highest amount of oxygen that patients can consume during incremental aerobic exercise and is considered the best indicator of exercise capacity.

SECONDARY OUTCOMES:
Double-product at the 11. minute of modified Bruce exercise test | From enrollment day to the end of the rehabilitation program at 4 weeks
  Double-product is obtained by multiplying heart rate and systolic blood pressure at a time point of exercise. It gradually increases as the workload increases during exercise. Double-product is an indirect indicator of myocardial oxygen demand. In this study a specific time point, 11. minute of the modified Bruce exercise test was addressed. There were two reasons for this. First, most patients pass the ventilatory anaerobic threshold between the 9. to 12. minutes of the modified Bruce testing protocol. The other reason is to compare the double product value at a similar workload before and after the rehabilitation program.
Oxygen (O₂) pulse at maximal exercise | From enrollment day to the end of the rehabilitation program at 4 weeks
  The oxygen pulse expresses the volume of oxygen expelled from the ventricles in each heartbeat. It is calculated by dividing the amount of oxygen consumed in one minute by the heart rate, that is, by the formula VO₂/heart rate. Its unit is expressed as ml/beat. This ratio is equal to the product of the stroke volume and the arteriovenous oxygen difference. Therefore, it reflects the change in stroke volume and the oxygen utilization capacity of the muscles during exercise.
Carbon dioxide respiratory equivalent (VE/VCO₂) | From enrollment day to the end of the rehabilitation program at 4 weeks
  The respiratory equivalent of carbon dioxide is expressed as VE/VCO₂ and is the ratio of the current minute ventilation (VE) to the carbon dioxide production (VCO₂) during incremental aerobic exercise. It is the amount of breathing required to remove the produced CO₂. It represents dead space ventilation and increases in patients with lung diseases such as heart failure and pulmonary hypertension.
Exercise time at which Ventilation Anaerobic Threshold (VAT) is reached | From enrollment day to the end of the rehabilitation program at 4 weeks
  The ventilatory anaerobic threshold (VAT) refers to the point during incremental exercise at which ventilation increases disproportionately to oxygen consumption (VO₂) due to a rise in carbon dioxide (CO₂) production. This marks the transition from predominantly aerobic metabolism, where oxygen is used to produce energy, to increased anaerobic metabolism, where the body starts relying more on non-oxygen-dependent processes for energy production.
  As exercise intensity increases, the muscles begin to produce more lactate. When the production of lactate exceeds the body's ability to clear it efficiently, it starts to accumulate in the bloodstream. To buffer the acid produced by lactate, the body produces more CO₂, leading to a corresponding increase in breathing rate (ventilation) to eliminate the excess CO₂. In this study, the time point to achieve VAT in the modified Bruce exercise test protocol was recorded.
First-Minute Heart Rate Recovery | From enrollment day to the end of the rehabilitation program at 4 weeks
  Heart rate recovery (HRR) refers to the rate at which the heart rate declines following the cessation of exercise, reflecting the balance of autonomic nervous system function, specifically the reactivation of parasympathetic (vagal) tone and withdrawal of sympathetic stimulation. In this study, HRR was assessed as the reduction in heart rate within the first minute of recovery after maximal exertion during exercise testing. A faster HRR is generally considered a marker of superior cardiovascular fitness and autonomic function. Conversely, impaired HRR, particularly a decline of fewer than 12 beats per minute in the first minute post-exercise, has been strongly associated with increased cardiovascular and all-cause mortality, as highlighted in numerous studies. This makes HRR a valuable prognostic tool in assessing long-term outcomes in patients with cardiovascular disease.
Fear of Activity in Patients With Coronary Artery Disease (Fact-CAD) score | From enrollment day to the end of the rehabilitation program at 4 weeks
  FACT-CAD is a scale used to measure fear of activity in patients with CAD. It consists of 21 questions that evaluate fear of activity and behavioural changes in patients with CAD. Each question receives an answer as ''always, often, sometimes, very rarely, never''. The data obtained allow us to comment on the patient's post-cardiac event behavioural changes and fear of activity. A higher score represents an increased fear of activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ülkü Nesrin Demirsoy, MD, Principal Investigator — Gazi University Faculty of Medicine; Nihan Burhandağ, MD, Principal Investigator — Gazi University Faculty of Medicine; Levent Karataş, MD, Principal Investigator — Gazi University Faculty of Medicine
Locations (1):
- Gazi University Hospital, Department of Physical Medicine and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kraal JJ, Peek N, Van den Akker-Van Marle ME, Kemps HM. Effects of home-based training with telemonitoring guidance in low to moderate risk patients entering cardiac rehabilitation: short-term results of the FIT@Home study. Eur J Prev Cardiol. 2014 Nov;21(2 Suppl):26-31. doi: 10.1177/2047487314552606. PMID 25354951
- [Background] Amaravathi E, Ramarao NH, Raghuram N, Pradhan B. Yoga-Based Postoperative Cardiac Rehabilitation Program for Improving Quality of Life and Stress Levels: Fifth-Year Follow-up through a Randomized Controlled Trial. Int J Yoga. 2018 Jan-Apr;11(1):44-52. doi: 10.4103/ijoy.IJOY_57_16. PMID 29343930
- [Background] Ozyemisci-Taskiran O, Demirsoy N, Atan T, Yuksel S, Coskun O, Aytur YK, Tur BS, Karakas M, Turak O, Topal S. Development and Validation of a Scale to Measure Fear of Activity in Patients With Coronary Artery Disease (Fact-CAD). Arch Phys Med Rehabil. 2020 Mar;101(3):479-486. doi: 10.1016/j.apmr.2019.09.001. Epub 2019 Sep 25. PMID 31562874
- [Background] WASSERMAN K, MCILROY MB. DETECTING THE THRESHOLD OF ANAEROBIC METABOLISM IN CARDIAC PATIENTS DURING EXERCISE. Am J Cardiol. 1964 Dec;14:844-52. doi: 10.1016/0002-9149(64)90012-8. No abstract available. PMID 14232808
- [Background] Forman DE, Myers J, Lavie CJ, Guazzi M, Celli B, Arena R. Cardiopulmonary exercise testing: relevant but underused. Postgrad Med. 2010 Nov;122(6):68-86. doi: 10.3810/pgm.2010.11.2225. PMID 21084784
- [Background] Holverda S, Bogaard HJ, Groepenhoff H, Postmus PE, Boonstra A, Vonk-Noordegraaf A. Cardiopulmonary exercise test characteristics in patients with chronic obstructive pulmonary disease and associated pulmonary hypertension. Respiration. 2008;76(2):160-7. doi: 10.1159/000110207. Epub 2007 Oct 25. PMID 17960052
- [Background] Albouaini K, Egred M, Alahmar A, Wright DJ. Cardiopulmonary exercise testing and its application. Postgrad Med J. 2007 Nov;83(985):675-82. doi: 10.1136/hrt.2007.121558. PMID 17989266
- [Background] Arena R, Myers J, Abella J, Peberdy MA, Bensimhon D, Chase P, Guazzi M. Development of a ventilatory classification system in patients with heart failure. Circulation. 2007 May 8;115(18):2410-7. doi: 10.1161/CIRCULATIONAHA.107.686576. Epub 2007 Apr 23. PMID 17452607
- [Background] Lauer M, Froelicher ES, Williams M, Kligfield P; American Heart Association Council on Clinical Cardiology, Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention. Exercise testing in asymptomatic adults: a statement for professionals from the American Heart Association Council on Clinical Cardiology, Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention. Circulation. 2005 Aug 2;112(5):771-6. doi: 10.1161/CIRCULATIONAHA.105.166543. Epub 2005 Jul 5. PMID 15998671
- [Background] Batalik L, Dosbaba F, Hartman M, Batalikova K, Spinar J. Benefits and effectiveness of using a wrist heart rate monitor as a telerehabilitation device in cardiac patients: A randomized controlled trial. Medicine (Baltimore). 2020 Mar;99(11):e19556. doi: 10.1097/MD.0000000000019556. PMID 32176113